CLINICAL TRIAL: NCT01167517
Title: Lactation Education Study in Mothers of Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Forsyth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00013359; FMC 2010.0401 (Other: Forsyth Medical Center)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-08

CONDITIONS: Infant, Very Low Birth Weight; Lactation
Keywords: Breast milk; Feeding; Prematurity; Low birth weight infant; Low maternal breast milk feeding
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructional digital video disc (DVD) (Experimental): Breast milk expression instructions provided by digital video disc at the time of hospital discharge.
  Interventions: Other: Instructional digital video disc (DVD)
- Instructions in print format (Placebo Comparator): Breast milk expression instructions provided in print format at the time of hospital discharge.
  Interventions: Other: Instructional digital video disc (DVD)

INTERVENTIONS:
Other: Instructional digital video disc (DVD) — Breast milk expression instructions provided by digital video disc at the time of hospital discharge
  Other Names: A Premie Needs His Mother

SUMMARY:
This study will test the effectiveness of breast milk expression discharge instructions in digital video disc (DVD) format for home use by mothers of very low birth weight infants on the dose and duration of mother's breast milk feeding in their infants compared to breast milk expression discharge instructions in printed format. The investigators hypothesize that infants whose mothers receive breast milk expression discharge instructions via DVD will receive a larger dose of maternal breast milk and for longer duration during the initial neonatal intensive care unit hospitalization than infants whose mothers receive discharge instructions in printed format.

DETAILED DESCRIPTION:
Very low birth weight (VLBW; <1500 g) infants who receive maternal breast milk, as opposed to infant formula, are less likely to experience the serious illnesses and poor developmental outcomes associated with VLBW. However, a disparity exists in breast milk feeding. Infants whose mothers have low educational attainment and low income are less likely to receive maternal breast milk than infants whose mothers who do not have low educational attainment and low income. The primary objective of this proposed research is to determine the effect of lactation discharge instructions in an audio-visual format provided to mothers for home viewing on the dose and duration of maternal breast milk received by their VLBW infants during the neonatal intensive care unit hospitalization.

Methods. Forty mothers of VLBW infants will be randomly assigned to receive a breast milk expression instruction digital video disc (DVD) in addition to standard of care lactation education or assigned to receive written instructions in addition to standard of care lactation education. In addition to comparing infant intake of maternal breast milk intake, pre and post intervention lactation and breast milk expression knowledge will be compared between groups and DVD viewing frequency and acceptability will be determined with a log and questionnaire to be completed by the intervention group and collected the first month after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Infant birth weight less than 1500 grams
* Maternal educational attainment less than/equal to 12 years
* Maternal low income status (Medicaid participant prior to delivery)

Exclusion Criteria:

* Non-English speaking
* Illicit drug use during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-04-09 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Maternal breast milk proportion of enteral feeding. | Daily during the initial hospitalization which is an average of 60 days
  Volume (ml) of maternal breast milk received daily by the infant divided by the total daily volume of all enteral feeding received.
Volume of daily maternal milk intake in relation to infant weight. | Daily during the initial hospitalization which is an average of 60 days
  Daily maternal milk intake(ml)divided by daily infant weight (kilograms).

SECONDARY OUTCOMES:
Maternal lactation and breast milk expression knowledge. | One month postpartum
  Prior knowledge will be assessed by administering a self-administered knowledge test on lactation and breast milk expression before providing the instructional DVD or written instructions. The same test will be self-administered approximately one month after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Sisk, PhD, Principal Investigator — Wake Forest Baptist Medical Center/ Forsyth Medical Center
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Ong J, Miller PS, Appleby R, Allegretto R, Gawlinski A. Effect of a preoperative instructional digital video disc on patient knowledge and preparedness for engaging in postoperative care activities. Nurs Clin North Am. 2009 Mar;44(1):103-15, xii. doi: 10.1016/j.cnur.2008.10.014. PMID 19167553
- [Background] Sisk PM, Lovelady CA, Dillard RG, Gruber KJ. Lactation counseling for mothers of very low birth weight infants: effect on maternal anxiety and infant intake of human milk. Pediatrics. 2006 Jan;117(1):e67-75. doi: 10.1542/peds.2005-0267. PMID 16396850
- [Background] Furman L, Taylor G, Minich N, Hack M. The effect of maternal milk on neonatal morbidity of very low-birth-weight infants. Arch Pediatr Adolesc Med. 2003 Jan;157(1):66-71. doi: 10.1001/archpedi.157.1.66. PMID 12517197
- [Background] Ronnestad A, Abrahamsen TG, Medbo S, Reigstad H, Lossius K, Kaaresen PI, Egeland T, Engelund IE, Irgens LM, Markestad T. Late-onset septicemia in a Norwegian national cohort of extremely premature infants receiving very early full human milk feeding. Pediatrics. 2005 Mar;115(3):e269-76. doi: 10.1542/peds.2004-1833. Epub 2005 Feb 1. PMID 15687416
- [Background] Schanler RJ, Hurst NM, Lau C. The use of human milk and breastfeeding in premature infants. Clin Perinatol. 1999 Jun;26(2):379-98, vii. PMID 10394493
- [Background] Schanler RJ, Shulman RJ, Lau C. Feeding strategies for premature infants: beneficial outcomes of feeding fortified human milk versus preterm formula. Pediatrics. 1999 Jun;103(6 Pt 1):1150-7. doi: 10.1542/peds.103.6.1150. PMID 10353922
- [Background] Sisk PM, Lovelady CA, Dillard RG, Gruber KJ, O'Shea TM. Early human milk feeding is associated with a lower risk of necrotizing enterocolitis in very low birth weight infants. J Perinatol. 2007 Jul;27(7):428-33. doi: 10.1038/sj.jp.7211758. Epub 2007 Apr 19. PMID 17443195
- [Background] Sisk PM, Lovelady CA, Gruber KJ, Dillard RG, O'Shea TM. Human milk consumption and full enteral feeding among infants who weigh </= 1250 grams. Pediatrics. 2008 Jun;121(6):e1528-33. doi: 10.1542/peds.2007-2110. PMID 18519456
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Background] Meier PP, Engstrom JL, Mingolelli SS, Miracle DJ, Kiesling S. The Rush Mothers' Milk Club: breastfeeding interventions for mothers with very-low-birth-weight infants. J Obstet Gynecol Neonatal Nurs. 2004 Mar-Apr;33(2):164-74. doi: 10.1177/0884217504263280. PMID 15095795
- [Background] Jones E, Spencer SA. Optimising the provision of human milk for preterm infants. Arch Dis Child Fetal Neonatal Ed. 2007 Jul;92(4):F236-8. doi: 10.1136/adc.2006.100941. PMID 17585091
- [Background] Killersreiter B, Grimmer I, Buhrer C, Dudenhausen JW, Obladen M. Early cessation of breast milk feeding in very low birthweight infants. Early Hum Dev. 2001 Jan;60(3):193-205. doi: 10.1016/s0378-3782(00)00116-x. PMID 11146238

DOCUMENTS (1):
  • Informed Consent Form (2010-01-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01167517/ICF_000.pdf